CLINICAL TRIAL: NCT00826514
Title: A PHASE 2, 16 WEEK, MULTICENTER, RANDOMIZED, DOUBLE-BLIND PLACEBO-CONTROLLED, PARALLEL GROUP PROOF-OF-CONCEPT STUDY EVALUATING THE EFFICACY AND SAFETY OF TANEZUMAB FOR THE TREATMENT OF PAIN ASSOCIATED WITH CHRONIC ABACTERIAL PROSTATITIS
Brief Title: An Efficacy And Safety Study Of Tanezumab For The Treatment Of Pain Associated With Chronic Abacterial Prostatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091019; 2008-004861-25 (EudraCT Number); PROSTATITIS POC (Other: Alias Study Number)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: Chronic Prostatis
MeSH Terms: conditions — Prostatitis | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tanezumab (Experimental)
  Interventions: Drug: Tanezumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tanezumab — Intravenous, 20 mg, single dose.
  Arms: Tanezumab
Drug: Placebo — Intravenous placebo, single dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether tanezumab is effective in the treatment of pain associated with chronic prostatitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic prostatitis
* Male adults at least 18 years of age
* Moderate to severe chronic prostatitis, with an average pain score above a pre-defined level
* To use contraception.

Exclusion Criteria:

* History of symptoms for less than 3 of the last 6 months
* History of recurrent urinary tract infections, or genito-urinary cancer
* Use of finasteride or dutasteride within 6 months.
* History of hepatitis B, C or human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 62 (Actual)
Dates: Start 2009-03-25 (Actual); Primary Completion 2010-01-11 (Actual); Study Completion 2010-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (23):
  - Alabama Research Center, LLC, Birmingham, Alabama
  - The Kirklin Clinic, Birmingham, Alabama
  - University of Alabama Birmingham, Birmingham, Alabama
  - Valley Urologic Associates, Goodyear, Arizona
  - Dedicated Clinical Research, Litchfield Park, Arizona
  - Clinical Innovations, Inc., Costa Mesa, California
  - Citrus Valley Medical Research Inc., Glendora, California
  - Atlantic Urological Medical Group Incorporated, Long Beach, California
  - Orange Coast Urology, Newport Beach, California
  - Los Angeles Infertility and Prostatitis Medical Group, Santa Monica, California
  - Specialists in Urology, Bonita Springs, Florida
  - Specialists in Urology, Naples, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - Regional Urology, LLC, Shreveport, Louisiana
  - Quality Clinical Research, Omaha, Nebraska
  - Hudson Valley Urology, PC, Kingston, New York
  - University Urology Associates, New York, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - Tri-State Urologic Services PSC, Inc. dba The Urology Group, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University of the Commonwealth System of Higher Education, Philadelphia, Pennsylvania
  - University Urology, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
- Canada (12):
  - Prostate Cancer Centre / Urology Research, Calgary, Alberta
  - Office of Dr. Nazmuddin Merali, Victoria, British Columbia
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - PJ Pommerville Inc., Victoria, British Columbia
  - Dr. Steinhoff Clinical Research, Victoria, British Columbia
  - Manitoba Prostate Centre, Winnipeg, Manitoba
  - The Male/Female Health and Research Centre, Barrie, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Centre for Applied Urological Research, Kingston, Ontario
  - Urology Associates / Urologic Medical Research, Kitchener, Ontario
  - The Male Health Centre, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
- France (5):
  - Hopital Edouard Herriot, Lyon
  - Centre Hospitalier Universitaire de NANTES (CHU), Nantes
  - CHU de Nîmes - Hôpital CAREMEAU, Nîmes
  - Hopital TENON, Paris
  - Hopital Rothschild, Paris
- Sweden (2):
  - Capio Citykliniken AB, Lund
  - Skaraborgs Sjukhus, FoU-centrum och urologkliniken, Skövde
- Switzerland (2):
  - Universitaetsspital Basel, Urologische Klinik, Basel
  - Klinik und Poliklinik fuer Urologie, Inselspital, Bern

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091019&StudyName=An%20Efficacy%20And%20Safety%20Study%20Of%20Tanezumab%20For%20The%20Treatment%20Of%20Pain%20Associated%20With%20Chronic%20Abacterial%20Prostatitis

RESULTS

PARTICIPANT FLOW:
Groups:
- Tanezumab: A single dose of tanezumab (RN624 or PF-04383119) 20 milligram (mg) intravenous infusion over 5 minutes. Participants were followed up to Week 16.
- Placebo: A single dose of placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion over 5 minutes. Participants were followed up to Week 16.
Period: Overall Study
Arm/Group | Tanezumab | Placebo
Started | 30 | 32
Completed | 27 | 27
Not Completed | 3 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 8 | 18 | 26
  45 to 64 years | 17 | 12 | 29
  Greater than or equal to (>=) 65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Pain Score at Week 6
Description: Participants assessed average chronic prostatitis pain in the last 24 hours on an 11-point numeric rating scale (NRS) ranging from 0 (no chronic prostatitis pain) to 10 (chronic prostatitis pain as bad as you can imagine). The average daily pain score was calculated as the mean of the scores over the last 7 days prior to each assessment time point. Higher score indicated severe pain.
Time Frame: Baseline, Week 6
Population: Restricted Full Analysis Set (rFAS): all randomized participants who received at least 1 treatment dose, completed at least 4 diary days during 7 day prior randomization, and had baseline, post-randomization primary efficacy data for 4 or more days within assessment window or for 2 or more consecutive days for diary endpoints derived from 3-day diary. Overall number of participants analyzed=participants evaluable for this measure; number analyzed=participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 31
units on a scale
  Baseline | 5.5 (1.10) | 5.6 (1.14)
  Change at Week 6: number analyzed (Participants) | 27 | 28
  Change at Week 6 | -1.4 (1.43) | -1.0 (1.43)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Analysis was based on analysis of co-variance (ANCOVA) model with baseline value, age and treatment as covariates; Test type: Superiority or Other; Least squares mean difference = -0.47, 95% CI 2-sided [-1.150 to 0.209], Standard Error of Mean 0.392

2. Secondary Outcome: Change From Baseline in Average Daily Pain Score at Weeks 2, 4, 8, 10, and 16
Description: as for outcome 1
Time Frame: Baseline, Weeks 2, 4, 8, 10, and 16
Population: Analysis was performed on rFAS. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale
  Change at Week 2 | -0.8 (1.43) | -1.1 (1.13)
  Change at Week 4: number analyzed (Participants) | 29 | 28
  Change at Week 4 | -1.6 (1.51) | -0.9 (1.37)
  Change at Week 8: number analyzed (Participants) | 26 | 24
  Change at Week 8 | -1.5 (1.46) | -1.3 (1.61)
  Change at Week 10: number analyzed (Participants) | 26 | 24
  Change at Week 10 | -1.5 (1.62) | -1.4 (1.58)
  Change at Week 16: number analyzed (Participants) | 15 | 12
  Change at Week 16 | -1.8 (1.30) | -1.9 (1.47)

3. Secondary Outcome: Change From Baseline in Worst Daily Pain Score at Weeks 2, 4, 6, 8, 10, and 16
Description: Participants assessed worst chronic prostatitis pain in the last 24 hours on an 11-point numeric rating scale (NRS) ranging from 0 (no chronic prostatitis pain) to 10 (chronic prostatitis pain as bad as you can imagine). The worst daily pain score was calculated as the mean of the scores over the last 7 days prior to each assessment time point. Higher score indicated severe pain.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 16
Population: Analysis was performed on rFAS. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' evaluable participants at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 31
units on a scale
  Baseline | 6.4 (1.17) | 6.8 (1.12)
  Change at Week 2: number analyzed (Participants) | 30 | 30
  Change at Week 2 | -0.7 (1.75) | -1.2 (1.31)
  Change at Week 4: number analyzed (Participants) | 29 | 28
  Change at Week 4 | -1.6 (1.85) | -0.9 (1.55)
  Change at Week 6: number analyzed (Participants) | 27 | 28
  Change at Week 6 | -1.4 (1.95) | -1.1 (1.43)
  Change at Week 8: number analyzed (Participants) | 26 | 24
  Change at Week 8 | -1.3 (2.01) | -1.4 (1.86)
  Change at Week 10: number analyzed (Participants) | 26 | 24
  Change at Week 10 | -1.4 (2.01) | -1.7 (1.82)
  Change at Week 16: number analyzed (Participants) | 15 | 12
  Change at Week 16 | -1.8 (1.79) | -2.1 (1.62)

4. Secondary Outcome: Change From Baseline in National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI) Overall and Sub-scale Score at Weeks 2, 4, 6, 8, 10, and 16
Description: CPSI is a 9-item questionnaire, contains 3 modules that measure pain (question 1 to 4), urinary symptoms (question 5 and 6) and global quality of life (question 7 to 9). Total scores range from 0 to 21 on the pain module, 0 to 10 on the urinary symptoms and 0 to 12 on the quality of life module. NIH-CPSI total score (9-items) range from 0 to 43. Higher total and module scores indicate greater symptom severity and bother.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 16
Population: Analysis was performed on rFAS. Here, 'number analyzed' signifies evaluable participants at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 32
units on a scale
  Baseline: CPSI Total Score | 25.5 (4.91) | 26.4 (4.38)
  Baseline: CPSI Pain Domain (PD) Score | 13.0 (2.09) | 13.5 (1.85)
  Baseline: CPSI Urinary Symptom (US) Score | 4.2 (2.39) | 4.1 (2.88)
  Baseline: CPSI Quality of Life (QoL) Score | 8.3 (2.18) | 8.8 (1.87)
  Change at Week 2: CPSI Total Score: number analyzed (Participants) | 27 | 28
  Change at Week 2: CPSI Total Score | -3.2 (6.72) | -3.1 (5.92)
  Change at Week 2: CPSI PD Score: number analyzed (Participants) | 27 | 28
  Change at Week 2: CPSI PD Score | -2.3 (3.44) | -1.8 (2.78)
  Change at Week 2: CPSI US Score: number analyzed (Participants) | 27 | 28
  Change at Week 2: CPSI US Score | 0.2 (2.25) | -0.3 (2.29)
  Change at Week 2: CPSI QoL Score: number analyzed (Participants) | 27 | 28
  Change at Week 2: CPSI QoL Score | -1.0 (2.47) | -1.0 (1.69)
  Change at Week 4: CPSI Total Score: number analyzed (Participants) | 25 | 27
  Change at Week 4: CPSI Total Score | -5.2 (6.56) | -3.5 (6.27)
  Change at Week 4: CPSI PD Score: number analyzed (Participants) | 25 | 27
  Change at Week 4: CPSI PD Score | -3.5 (3.63) | -2.0 (2.72)
  Change at Week 4: CPSI US Score: number analyzed (Participants) | 25 | 27
  Change at Week 4: CPSI US Score | 0.1 (2.44) | -0.7 (2.80)
  Change at Week 4: CPSI QoL Score: number analyzed (Participants) | 25 | 27
  Change at Week 4: CPSI QoL Score | -1.8 (2.71) | -0.9 (1.96)
  Change at Week 6: CPSI Total Score: number analyzed (Participants) | 25 | 26
  Change at Week 6: CPSI Total Score | -4.3 (7.04) | -4.0 (7.06)
  Change at Week 6: CPSI PD Score: number analyzed (Participants) | 25 | 26
  Change at Week 6: CPSI PD Score | -2.8 (3.64) | -2.2 (2.94)
  Change at Week 6: CPSI US Score: number analyzed (Participants) | 25 | 26
  Change at Week 6: CPSI US Score | -0.2 (2.38) | -0.8 (3.18)
  Change at Week 6: CPSI QoL Score: number analyzed (Participants) | 25 | 26
  Change at Week 6: CPSI QoL Score | -1.3 (2.67) | -1.0 (2.32)
  Change at Week 8: CPSI Total Score: number analyzed (Participants) | 25 | 24
  Change at Week 8: CPSI Total Score | -3.0 (5.73) | -4.8 (7.55)
  Change at Week 8: CPSI PD Score: number analyzed (Participants) | 25 | 24
  Change at Week 8: CPSI PD Score | -2.1 (3.15) | -2.9 (3.97)
  Change at Week 8: CPSI US Score: number analyzed (Participants) | 25 | 24
  Change at Week 8: CPSI US Score | -0.0 (1.72) | -0.5 (2.65)
  Change at Week 8: CPSI QoL Score: number analyzed (Participants) | 25 | 24
  Change at Week 8: CPSI QoL Score | -0.8 (2.36) | -1.4 (2.48)
  Change at Week 10: CPSI Total Score: number analyzed (Participants) | 21 | 26
  Change at Week 10: CPSI Total Score | -2.9 (6.06) | -4.9 (7.62)
  Change at Week 10: CPSI PD Score: number analyzed (Participants) | 21 | 26
  Change at Week 10: CPSI PD Score | -2.4 (3.56) | -3.0 (3.64)
  Change at Week 10: CPSI US Score: number analyzed (Participants) | 21 | 26
  Change at Week 10: CPSI US Score | 0.6 (1.96) | -0.7 (2.59)
  Change at Week 10: CPSI QoL Score: number analyzed (Participants) | 21 | 26
  Change at Week 10: CPSI QoL Score | -1.1 (2.20) | -1.2 (2.87)
  Change at Week 16: CPSI Total Score: number analyzed (Participants) | 23 | 22
  Change at Week 16: CPSI Total Score | -4.0 (6.34) | -5.3 (7.62)
  Change at Week 16: CPSI PD Score: number analyzed (Participants) | 23 | 22
  Change at Week 16: CPSI PD Score | -2.4 (3.06) | -3.2 (3.93)
  Change at Week 16: CPSI US Score: number analyzed (Participants) | 23 | 22
  Change at Week 16: CPSI US Score | -0.3 (2.08) | -0.5 (2.76)
  Change at Week 16: CPSI QoL Score: number analyzed (Participants) | 23 | 22
  Change at Week 16: CPSI QoL Score | -1.2 (2.35) | -1.6 (2.59)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Change at Week 6, CPSI Total Score: Analysis was based on ANCOVA model with baseline value, age, baseline pain stratification group and treatment as covariates; Test type: Superiority or Other; Least squares mean difference = -1.42, 90% CI 2-sided [-4.754 to 1.905], Standard Error of Mean 1.901
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Change at Week 6, CPSI PD Score: Analysis was based on ANCOVA model with baseline value, age, baseline pain stratification group and treatment as covariates; Test type: Superiority or Other; Least squares mean difference = -1.06, 90% CI 2-sided [-2.701 to 0.591], Standard Error of Mean 0.931
Statistical Analysis 3: Comparison: Tanezumab vs Placebo; Change at Week 6, CPSI US Score: Analysis was based on ANCOVA model with baseline value, age, baseline pain stratification group and treatment as covariates; Test type: Superiority or Other; Least squares mean difference = 0.38, 90% CI 2-sided [-0.789 to 1.541], Standard Error of Mean 0.670
Statistical Analysis 4: Comparison: Tanezumab vs Placebo; Change at Week 6, CPSI QoL Score: Analysis was based on ANCOVA model with baseline value, age, baseline pain stratification group and treatment as covariates; Test type: Superiority or Other; Least squares mean difference = -0.58, 90% CI 2-sided [-1.785 to 0.631], Standard Error of Mean 0.697

5. Secondary Outcome: Change From Baseline in Number of Micturitions Per 24 Hours at Weeks 2, 4, 6, 8, 10, and 16
Description: The micturition frequency per 24 hours was calculated from the sum of voluntary voids divided by the diary period over which they were collected.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 24 | 27
micturitions per 24 hours
  Baseline | 9.1 (3.70) | 9.4 (4.75)
  Change at Week 2: number analyzed (Participants) | 23 | 25
  Change at Week 2 | 0.9 (2.86) | -0.3 (3.32)
  Change at Week 4: number analyzed (Participants) | 21 | 21
  Change at Week 4 | 0.3 (2.45) | -0.6 (4.10)
  Change at Week 6: number analyzed (Participants) | 23 | 26
  Change at Week 6 | 0.3 (1.92) | -0.3 (3.54)
  Change at Week 8: number analyzed (Participants) | 18 | 19
  Change at Week 8 | 0.6 (3.50) | -0.7 (4.69)
  Change at Week 10: number analyzed (Participants) | 21 | 21
  Change at Week 10 | 1.0 (2.92) | -1.2 (3.76)
  Change at Week 16: number analyzed (Participants) | 20 | 22
  Change at Week 16 | 0.3 (1.96) | -0.8 (4.25)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Change at Week 6: Analysis was based on ANCOVA model with baseline value, age, baseline pain stratification group and treatment as covariates; Test type: Superiority or Other; Least squares mean difference = 0.18, 90% CI 2-sided [-0.990 to 1.348], Standard Error of Mean 0.649

6. Secondary Outcome: Change From Baseline in Number of Nocturnal Micturitions Per 24 Hours at Weeks 2, 4, 6, 8, 10, and 16
Description: Nocturnal micturition was calculated as the sum of voluntary voids that occur during a night's sleep, divided by the number of nights over which this was collected.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 16
Population: Analysis was performed on rFAS. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number anlayzed' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 24 | 25
micturitions per 24 hours
  Baseline | 3.0 (3.24) | 3.8 (3.56)
  Change at Week 2: number analyzed (Participants) | 23 | 23
  Change at Week 2 | -0.2 (2.45) | -1.2 (3.43)
  Change at Week 4: number analyzed (Participants) | 21 | 20
  Change at Week 4 | -0.6 (3.09) | -1.2 (2.65)
  Change at Week 6: number analyzed (Participants) | 23 | 23
  Change at Week 6 | -0.4 (3.45) | -0.8 (3.91)
  Change at Week 8: number analyzed (Participants) | 18 | 17
  Change at Week 8 | 0.9 (3.39) | 0.4 (3.30)
  Change at Week 10: number analyzed (Participants) | 21 | 19
  Change at Week 10 | -1.0 (2.77) | -0.6 (3.39)
  Change at Week 16: number analyzed (Participants) | 19 | 20
  Change at Week 16 | -0.8 (1.48) | -1.4 (3.89)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least squares mean difference = -0.19, 90% CI 2-sided [-1.829 to 1.452], Standard Error of Mean 0.930

7. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition at Weeks 2, 4, 6, 8, 10, and 16
Description: Mean voided volume per micturition was calculated as the total urine volume voided (resulting from a toilet [voluntary] void) during the diary period when this was measured, divided by the number of toilet voids over which this occurred.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 24 | 27
milliliter
  Baseline | 216.7 (90.04) | 208.5 (86.38)
  Change at Week 2: number analyzed (Participants) | 23 | 25
  Change at Week 2 | -13.8 (47.95) | 26.8 (66.13)
  Change at Week 4: number analyzed (Participants) | 21 | 21
  Change at Week 4 | -17.4 (46.49) | 12.1 (62.80)
  Change at Week 6: number analyzed (Participants) | 23 | 26
  Change at Week 6 | -24.7 (58.94) | 8.3 (68.48)
  Change at Week 8: number analyzed (Participants) | 17 | 19
  Change at Week 8 | -7.4 (48.11) | 11.0 (68.07)
  Change at Week 10: number analyzed (Participants) | 21 | 21
  Change at Week 10 | -27.5 (63.45) | 20.3 (74.81)
  Change at Week 16: number analyzed (Participants) | 20 | 22
  Change at Week 16 | -27.4 (48.32) | 15.0 (67.92)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least squares mean difference = -33.56, 90% CI 2-sided [-64.144 to -2.968], Standard Error of Mean 17.026

8. Secondary Outcome: Change From Baseline in Mean Urinary Event Pain Score Per 24 Hours at Weeks 2, 4, 6, 8, 10, and 16
Description: Subject assessed discrete urinary events: voluntary toilet voids (with volume voided), and urgency episodes. For each urinary event, subjects assessed the level of pain intensity on a 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Mean pain severity per urinary event (toilet void, urgency episode) was calculated as the mean of all pain severities over the last 7 days prior to each assessment time point. Higher score indicated severe pain.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 24 | 27
units on a scale
  Baseline | 3.0 (2.37) | 3.6 (1.99)
  Change at Week 2: number analyzed (Participants) | 23 | 25
  Change at Week 2 | -0.2 (1.39) | -0.4 (1.29)
  Change at Week 4: number analyzed (Participants) | 21 | 21
  Change at Week 4 | -0.7 (1.41) | -0.5 (1.55)
  Change at Week 6: number analyzed (Participants) | 23 | 26
  Change at Week 6 | -0.6 (1.37) | -0.3 (2.03)
  Change at Week 8: number analyzed (Participants) | 17 | 19
  Change at Week 8 | -0.7 (1.49) | -0.6 (1.88)
  Change at Week 10: number analyzed (Participants) | 21 | 21
  Change at Week 10 | -0.6 (1.32) | -1.0 (1.59)
  Change at Week 16: number analyzed (Participants) | 20 | 22
  Change at Week 16 | -0.7 (1.34) | -0.8 (2.04)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least squares mean difference = -0.47, 90% CI 2-sided [-1.364 to 0.415], Standard Error of Mean 0.489

9. Secondary Outcome: Change From Baseline in Urinary Urgency Episodes Per 24 Hours at Weeks 2, 4, 6, 8, 10, and 16
Description: Urinary urgency episodes per 24 hours was calculated as the sum of any urgency episodes occurring during the diary period when this was measured, divided by the number of days over which they were recorded.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: urgency episodes per 24 hours
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 24 | 27
urgency episodes per 24 hours
  Baseline | 4.7 (5.65) | 5.1 (5.50)
  Change at Week 2: number analyzed (Participants) | 23 | 25
  Change at Week 2 | 0.3 (3.14) | -0.3 (4.08)
  Change at Week 4: number analyzed (Participants) | 21 | 21
  Change at Week 4 | -0.9 (3.03) | 0.2 (5.10)
  Change at Week 6: number analyzed (Participants) | 23 | 26
  Change at Week 6 | -0.8 (1.44) | 0.0 (4.90)
  Change at Week 8: number analyzed (Participants) | 18 | 19
  Change at Week 8 | 0.3 (3.59) | 0.6 (5.86)
  Change at Week 10: number analyzed (Participants) | 21 | 21
  Change at Week 10 | -0.1 (3.58) | -0.7 (5.67)
  Change at Week 16: number analyzed (Participants) | 20 | 22
  Change at Week 16 | -1.4 (2.25) | -0.6 (5.35)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least squares mean difference = -1.37, 90% CI 2-sided [-3.146 to 0.401], Standard Error of Mean 0.990

10. Secondary Outcome: Change From Baseline in Mean Sleep Disturbance Score Per 24 Hours at Weeks 2, 4, 6, 8, 10, and 16
Description: Mean sleep disturbance score was calculated from the sleep disturbance experienced over the previous night. The average sleep disturbance score per night was determined from calculating an average of all sleep disturbance scores in the 7 days prior to each assessment time point. Participants answered: "Over the past 24 hours, how much did the symptoms that you associate with your chronic prostatitis disturb your sleep?" Participants responded on a 5-points rating scale, ranged from 0 = not at all, 1 = a little, 2 = somewhat, 3 = very, and 4 = extremely. Higher score indicated greater sleep disturbance.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 16
Population: Analysis was performed on rFAS. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and number analyzed' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 31
units on a scale
  Baseline | 1.9 (0.80) | 1.7 (1.00)
  Change at Week 2: number analyzed (Participants) | 30 | 30
  Change at Week 2 | -0.3 (0.93) | -0.4 (0.54)
  Change at Week 4: number analyzed (Participants) | 29 | 28
  Change at Week 4 | -0.5 (0.79) | -0.3 (0.74)
  Change at Week 6: number analyzed (Participants) | 27 | 28
  Change at Week 6 | -0.4 (0.88) | -0.3 (0.75)
  Change at Week 8: number analyzed (Participants) | 26 | 24
  Change at Week 8 | -0.4 (0.91) | -0.4 (0.79)
  Change at Week 10: number analyzed (Participants) | 26 | 24
  Change at Week 10 | -0.4 (0.93) | -0.3 (0.82)
  Change at Week 16: number analyzed (Participants) | 15 | 12
  Change at Week 16 | -0.4 (0.81) | -0.4 (0.84)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least squares mean difference = -0.04, 90% CI 2-sided [-0.417 to 0.334], Standard Error of Mean 0.217

11. Secondary Outcome: Change From Baseline in Mean Pain Score Associated With Ejaculation Per 24 Hours at Weeks 2, 4, 6, 8, 10, and 16
Description: The participants were first asked whether they had ejaculated during the past 24 hours. If yes, they recorded how much pain related to ejaculation they had experienced during the past 24 hours by choosing the appropriate number an 11-point numeric rating scale (NRS) ranging from 0 (no ejaculatory pain at all) to 10 (ejaculatory pain as bad as you can imagine). Higher score indicated greater pain. Mean pain score associated with ejaculation was calculated from all ejaculation pain scores recorded in the 7 days prior to each assessment time point.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 17 | 19
units on a scale
  Baseline | 3.8 (2.40) | 3.4 (2.50)
  Change at Week 2: number analyzed (Participants) | 14 | 14
  Change at Week 2 | 0.3 (2.47) | -0.9 (1.37)
  Change at Week 4: number analyzed (Participants) | 14 | 13
  Change at Week 4 | -1.3 (1.30) | -0.3 (1.87)
  Change at Week 6: number analyzed (Participants) | 13 | 10
  Change at Week 6 | -1.5 (2.01) | -0.5 (1.69)
  Change at Week 8: number analyzed (Participants) | 13 | 12
  Change at Week 8 | -0.4 (1.94) | -0.4 (1.59)
  Change at Week 10: number analyzed (Participants) | 13 | 11
  Change at Week 10 | -1.0 (2.25) | -0.7 (1.68)
  Change at Week 16: number analyzed (Participants) | 6 | 5
  Change at Week 16 | -1.3 (1.76) | -1.6 (1.64)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least squares mean difference = 0.02, 90% CI 2-sided [-1.791 to 1.822], Standard Error of Mean 0.765

12. Secondary Outcome: Number of Participants With Global Response Assessment (GRA)
Description: The GRA questionnaire is a 7-point symmetric scale, which measured patient-reported overall response to treatment compared to baseline with the following possible responses: 1= markedly worse, 2 = moderately worse, 3= slightly worse, 4= no change, 5 = slightly improved,6 = moderately improved, and 7 = markedly improved. Participants who reported either of the latter 2 categories were defined as treatment responders. Participants were asked "Compared to when you began this trial, how would you rate your chronic prostatitis symptoms now?". Participants responded on 7-point symmetric scale ranged 1 to 7, where higher score indicated improvement.
Time Frame: Week 6 and 16
Population: Analysis was performed on rFAS. Here, 'overall number of participants analyzed) signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 25 | 26
Participants
  Week 6: Markedly Worse | 0 | 1
  Week 6: Moderately Worse | 2 | 1
  Week 6: Slightly Worse | 1 | 0
  Week 6: No Change | 6 | 11
  Week 6: Slightly Improved | 10 | 7
  Week 6: Moderately Improved | 3 | 5
  Week 6: Markedly Improved | 3 | 1
  Week 16: Markedly Worse: number analyzed (Participants) | 23 | 21
  Week 16: Markedly Worse | 0 | 0
  Week 16: Moderately Worse: number analyzed (Participants) | 23 | 21
  Week 16: Moderately Worse | 0 | 0
  Week 16: Slightly Worse: number analyzed (Participants) | 23 | 21
  Week 16: Slightly Worse | 1 | 0
  Week 16: No Change: number analyzed (Participants) | 23 | 21
  Week 16: No Change | 9 | 8
  Week 16: Slightly Improved: number analyzed (Participants) | 23 | 21
  Week 16: Slightly Improved | 8 | 6
  Week 16: Moderately Improved: number analyzed (Participants) | 23 | 21
  Week 16: Moderately Improved | 4 | 6
  Week 16: Markedly Improved: number analyzed (Participants) | 23 | 21
  Week 16: Markedly Improved | 1 | 1
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; Week 6: Logistic regression model with age, baseline pain stratification group and treatment as covariates; Test type: Superiority or Other; Odds Ratio (OR) = 1.833, 90% CI 2-sided [0.763 to 4.407]
Statistical Analysis 2: Comparison: Tanezumab vs Placebo; Week 16: Logistic regression model with age, baseline pain stratification group and treatment as covariates; Test type: Superiority or Other; Odds Ratio (OR) = 1.000, 90% CI 2-sided [0.388 to 2.575]

13. Secondary Outcome: Patient Global Satisfaction Assessment
Description: Participant global satisfaction was assessed using Patient Reported Treatment Impact (PRTI) which was a self-administered questionnaire containing four items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participant's answered the question "Overall, how satisfied are you with the drug that you received since you entered this trial?". Participants provided response on a 5-point scale where 1=extremely dissatisfied, 2=dissatisfied, 3=neither satisfied nor dissatisfied, 4=satisfied and 5=extremely satisfied. Higher score indicated greater satisfaction, preference or willingness to use study medication. Number of participants with each response is reported.
Time Frame: Week 6 and 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 25 | 24
Participants
  Week 6: Extremely Satisfied | 3 | 0
  Week 6: Satisfied | 5 | 5
  Week 6:Neither Satisfied nor Dissatisfied | 10 | 13
  Week 6: Dissatisfied | 5 | 3
  Week 6: Extremely Dissatisfied | 2 | 3
  Week 16: Extremely Satisfied: number analyzed (Participants) | 23 | 22
  Week 16: Extremely Satisfied | 4 | 1
  Week 16: Satisfied: number analyzed (Participants) | 23 | 22
  Week 16: Satisfied | 7 | 11
  Week16:Neither Satisfied nor Dissatisfied: number analyzed (Participants) | 23 | 22
  Week16:Neither Satisfied nor Dissatisfied | 5 | 7
  Week 16: Dissatisfied: number analyzed (Participants) | 23 | 22
  Week 16: Dissatisfied | 5 | 1
  Week 16: Extremely Dissatisfied: number analyzed (Participants) | 23 | 22
  Week 16: Extremely Dissatisfied | 2 | 2

14. Secondary Outcome: Participant Global Preference
Description: Participant global preference is assessed using PRTI which is a self-administered questionnaire containing four items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participant reported previous treatment under following categories: lifestyle interventions, physical therapies, training programs, drug treatment - taken by mouth, surgery or other prostate procedure (e.g, microwave treatment), and no treatment. Participant preference was assessed using following categories: definitely prefer study medication, slightly prefer study medication, no preference, slightly prefer previous treatment, and definitely prefer previous treatment. Number of participants under each of the categories is reported. For previous treatment, a single participant may be represented in more than 1 category.
Time Frame: Week 6 and 16
Population: Analysis was performed on rFAS. Here, ''overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 25 | 24
Participants
  Week 6: Lifestyle Interventions | 5 | 5
  Week 6: Physical Therapies | 2 | 4
  Week 6: Training Programs | 2 | 0
  Week 6:Drug treatment-taken by mouth | 19 | 14
  Week 6: Surgery/other prostate procedure | 0 | 2
  Week 6: No Treatment | 6 | 4
  Week 6: Definitely Prefer Current Drug | 4 | 5
  Week 6: Slight Preference for Current Drug | 7 | 5
  Week 6: No Preference | 13 | 12
  Week 6: Slight Preference, Prior Treatment | 0 | 0
  Week 6: Definitely Prefer Prior Treatment | 1 | 2
  Week 16: Lifestyle Interventions: number analyzed (Participants) | 23 | 22
  Week 16: Lifestyle Interventions | 7 | 7
  Week 16: Physical Therapies: number analyzed (Participants) | 23 | 22
  Week 16: Physical Therapies | 3 | 4
  Week 16: Training Programs: number analyzed (Participants) | 23 | 22
  Week 16: Training Programs | 3 | 3
  Week 16: Drug treatment-taken by mouth: number analyzed (Participants) | 23 | 22
  Week 16: Drug treatment-taken by mouth | 17 | 18
  Week 16: Surgery/other prostate procedure: number analyzed (Participants) | 23 | 22
  Week 16: Surgery/other prostate procedure | 1 | 0
  Week 16: No Treatment: number analyzed (Participants) | 23 | 22
  Week 16: No Treatment | 3 | 1
  Week 16: Definitely Prefer Current Drug: number analyzed (Participants) | 23 | 22
  Week 16: Definitely Prefer Current Drug | 9 | 8
  Week 16: Slight Preference for Current Drug: number analyzed (Participants) | 23 | 22
  Week 16: Slight Preference for Current Drug | 4 | 5
  Week 16: No Preference: number analyzed (Participants) | 23 | 22
  Week 16: No Preference | 8 | 6
  Week 16: Slight Preference, Prior Treatment: number analyzed (Participants) | 23 | 22
  Week 16: Slight Preference, Prior Treatment | 0 | 0
  Week 16: Definitely Prefer Prior Treatment: number analyzed (Participants) | 23 | 22
  Week 16: Definitely Prefer Prior Treatment | 2 | 3

15. Secondary Outcome: Patient Willingness to Re-use Medicine
Description: Participant willingness to re-use study medication was assessed using PRTI which is a self-administered questionnaire containing four items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participant willingness to re-use study medication was assessed using following categories: definitely want to re-use, might want to re-use, not sure, might not want to re-use, definitely would not want to re-use.
Time Frame: Week 6 and 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 25 | 24
Participants
  Week 6: Definitely Want | 6 | 8
  Week 6: Might Want | 6 | 4
  Week 6: Not Sure | 8 | 9
  Week 6: Might not Want | 2 | 0
  Week 6: Definitely Would not Want | 3 | 3
  Week 16: Definitely Want: number analyzed (Participants) | 23 | 22
  Week 16: Definitely Want | 10 | 11
  Week 16: Might Want: number analyzed (Participants) | 23 | 22
  Week 16: Might Want | 3 | 7
  Week 16: Not Sure: number analyzed (Participants) | 23 | 22
  Week 16: Not Sure | 4 | 1
  Week 16: Might not Want: number analyzed (Participants) | 23 | 22
  Week 16: Might not Want | 3 | 0
  Week 16: Definitely Would not Want: number analyzed (Participants) | 23 | 22
  Week 16: Definitely Would not Want | 3 | 3

16. Secondary Outcome: Percentage of Participants Who Received Rescue Medication
Description: In the event of inadequate pain relief or worsening symptoms of chronic prostatitis, participants were allowed to take acetaminophen/paracetamol 500 mg, tablets or capsules as rescue medication.
Time Frame: Weeks 2, 4, 6, 8, 10, and 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 32
percentage of participants
  Week 2 | 22 | 19
  Week 4 | 17 | 17
  Week 6 | 15 | 16
  Week 8 | 14 | 12
  Week 10 | 13 | 11
  Week 16 | 12 | 4

17. Secondary Outcome: Amount of Rescue Medication Taken
Description: as for outcome 16
Time Frame: Weeks 2, 4, 6, 8, 10, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram/week
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 22 | 19
milligram/week
  Week 2 | 2681.82 (1949.03) | 2289.47 (2110.26)
  Week 4: number analyzed (Participants) | 17 | 17
  Week 4 | 3117.65 (1833.11) | 2764.71 (1977.35)
  Week 6: number analyzed (Participants) | 15 | 16
  Week 6 | 3366.67 (2133.63) | 2281.25 (1923.27)
  Week 8: number analyzed (Participants) | 14 | 12
  Week 8 | 3500.00 (1605.28) | 2375.00 (1693.91)
  Week 10: number analyzed (Participants) | 13 | 11
  Week 10 | 4000.00 (2500.00) | 3363.64 (2916.26)
  Week 16: number analyzed (Participants) | 12 | 4
  Week 16 | 2208.33 (1630.09) | 1375.00 (1436.14)

18. Secondary Outcome: Serum and Urine Nerve Growth Factor (NGF) Levels
Description: Serum NGF level was measured using Immunoaffinity High Performance Liquid Chromatography - Tandem Mass spectrometry (HPLC-MS/MS).
Time Frame: Day 1 (1 hour pre-dose), Weeks 2, 6, 10, and 16
Population: FAS: all randomized participants who received at least 1 dose of treatment and completed at least 4 diary days during 7 days prior to randomization. Here, 'overall number of participants analyzed' signifies participants evaluable for this measure and 'number analyzed' participants evaluable at specified time point for each arm. Urine NGF levels not analyzed as reliable assay for measurement in urine could not be identified.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 30
picogram per milliliter (pg/mL)
  Serum NGF: Day 1: number analyzed (Participants) | 27 | 30
  Serum NGF: Day 1 | 31.1 (8.8) | 33.2 (8.4)
  Serum NGF: Week 2: number analyzed (Participants) | 27 | 27
  Serum NGF: Week 2 | 2750 (583) | 40.2 (12.8)
  Serum NGF: Week 6: number analyzed (Participants) | 24 | 27
  Serum NGF: Week 6 | 3909 (768) | 37.7 (11.0)
  Serum NGF: Week 10: number analyzed (Participants) | 25 | 21
  Serum NGF: Week 10 | 3840 (925) | 34.8 (12.4)
  Serum NGF: Week 16: number analyzed (Participants) | 30 | 28
  Serum NGF: Week 16 | 3025 (1224) | 35.3 (11.0)

19. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study medication and up to Week 16 that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 32
Participants
  AEs | 24 | 21
  SAEs | 1 | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Neurological Examination Abnormalities
Description: A neurological examination assessed the strength of groups of muscles of the head and neck, upper limbs and lower limbs, deep tendon reflexes and sensation (tactile, vibration, joint position sense and pin prick) of index fingers and great toes.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 32
Participants | 3 | 1

21. Secondary Outcome: Post-void Residual (PVR) Volume
Description: PVR volume, an objective assessment of the amount of urine left in the bladder after normal urination and was monitored whether the active treatment had an adverse effect on lower urinary tract voiding function. The PVR volume was assessed using trans-abdominal ultrasound (e.g., bladder scanner) with the participant in a supine position immediately after voluntary urination.
Time Frame: Baseline, Weeks 2, 6, and 16
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study treatment. Here, 'number analyzed' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Tanezumab | Placebo
Number analyzed (Participants) | 30 | 32
milliliter
  Baseline | 34.1 (38.87) | 33.8 (40.87)
  Week 2: number analyzed (Participants) | 28 | 30
  Week 2 | 19.6 (34.11) | 23.2 (36.18)
  Week 6: number analyzed (Participants) | 29 | 29
  Week 6 | 31.4 (46.74) | 23.4 (41.38)
  Week 16: number analyzed (Participants) | 29 | 30
  Week 16 | 26.4 (23.60) | 22.5 (26.61)

22. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 1 (1 hour pre-dose), Weeks 2, 6, and 16
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study treatment. Here 'number analyzed' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab
Number analyzed (Participants) | 30
Participants
  Day 1 | 0
  Week 2: number analyzed (Participants) | 25
  Week 2 | 0
  Week 6: number analyzed (Participants) | 27
  Week 6 | 0
  Week 16: number analyzed (Participants) | 28
  Week 16 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Tanezumab | Placebo
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/32
Other Adverse Events (participants affected / at risk) | 23/30 | 21/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=30) | Placebo (N=32)
Device breakage (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=30) | Placebo (N=32)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Injury associated with device (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Therapeutic response unexpected (General disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Semen analysis abnormal (Investigations) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Ligament pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Allodynia (Nervous system disorders) | 4 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3
Dysaesthesia (Nervous system disorders) | 1 | 0
Formication (Nervous system disorders) | 0 | 1
Head discomfort (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 2
Hyperaesthesia (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hyporeflexia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 8 | 2
Presyncope (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Prostatic pain (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 0
Peripheral coldness (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.